CLINICAL TRIAL: NCT02558998
Title: Improving Clinical Trial Awareness in NSCLC: Pilot Testing A Novel Healthcare IT Platform for Incorporating Education at the Point of Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UPCC 34514
Record Dates: First submitted 2015-06-19; First posted 2015-09-24 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Non-Small Cell Lung Carcinoma (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Survey

SUMMARY:
The objective of this study is to 1) evaluate the impact of a novel individualized care planning/ educational technology (the On Q Care Planning System or CPS) on oncology patient and provider knowledge, attitudes and beliefs about Non-Small Cell Lung Carcinoma (NSCLC) clinical trials, as well as 2) to evaluate the impact of the On Q CPS on patient referral to and enrollment in NSCLC clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be 18 years of age or older.
* Patient participants must have Stage III, IV and/or recurrent NSCLC.
* Patient participants must be at a point of treatment initiation/change or evaluation for treatment initiation/change
* Patients must have working email address and internet access

Exclusion Criteria:

* Any participant who cannot understand written or spoken English.
* Any participant who is not competent to provide informed consent for study participation per the investigator.
* Any participant who cannot be present for the related study visits and/or complete the post-test assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-03; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Number of patient who completed surveys | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Bauml, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States